CLINICAL TRIAL: NCT05409196
Title: Phase 1 Two Stage Randomized, Double-blind, Placebo Controlled Dose- and Schedule Ranging Trial to Assess the Acute Safety, Tolerability, and Immunogenicity of a Live, Attenuated Shigella/ETEC Combination Vaccine Delivered Orally to Healthy Adults Age 18 to 45 Years Old
Brief Title: Phase 1 Trial for Safety, Tolerability, and Immunogenicity of a Live, Attenuated, Oral Shigella/ETEC Combination Vaccine to Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eveliqure Biotechnologies GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Prevention
Other Study IDs: EVQ 101
Record Dates: First submitted 2021-10-18; First posted 2022-06-08 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: Diarrheal Disease, Infectious; Gastrointestinal Disease; Reactive Arthritis
Keywords: Shigellosis
MeSH Terms: conditions — Dysentery; Gastrointestinal Diseases; Arthritis, Reactive; Dysentery, Bacillary | interventions — Vaccines

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ShigETEC vaccine (Experimental): In Stage 1 subjects will be allocated randomly to one of four study cohorts to receive a single oral dose of one of four escalating dose levels of ShigETEC vaccine (ShigETEC 1x10^9 CFU, ShigETEC 1x10^10 CFU, ShigETEC 5x10^10 CFU, ShigETEC 2x10^11 CFU). 8 subjects per dose group will be administered.
  Subjects in Stage 2 will be enrolled sequentially by group and allocated randomly to one of three study cohorts determined from Stage 1 to receive either two, three or four doses of the 5x10^10 ShigETEC vaccine at 3-day interval. 8 subjects per dose group will be administered.
  Interventions: Biological: ShigETEC live, attenuated, oral vaccine
- Placebo (Placebo Comparator): In Stage 1: 4 subjects in each dose group will receive a single oral dose of placebo
  In Stage 2: 4 subjects in each cohort will either receive 2, 3 or 4 doses of placebo at 3-day intervals.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: ShigETEC live, attenuated, oral vaccine — Vaccine or placebo will be delivered orally as a single dose in Stage 1 and between 2 and 4 doses at 3-day intervals in Stage 2 of the Study.
  Arms: ShigETEC vaccine
Drug: Placebo — Vaccine or placebo will be delivered orally as a single dose in Stage 1 and between 2 and 4 doses at 3-day intervals in Stage 2 of the Study.
  Arms: Placebo

SUMMARY:
This is a Phase 1 dose escalating study to assess the safety, tolerability, and immunogenicity of ShigETEC, a live, attenuated Shigella/ETEC combination vaccine given orally to healthy European adults 18 to 45 years of age.

The major aim is the development of an efficacious and safe vaccine that prevents diarrhea caused by Shigella and ETEC in travelers, military personal visiting endemic countries and children of the developing world.

This Phase 1 safety and immunogenicity study used a double-blind, placebo-control design and was conducted in two stages, a single ascending and a multiple ascending stage.

DETAILED DESCRIPTION:
ShigETEC vaccine is intended to stimulate an immune response in which protective antibodies are generated that prevent infection if a vaccinee is subsequently exposed to Shigella and ETEC.

Main objective of the study:

In Stage 1 is to determine Maximum Tolerated Single Dose of ShigETEC vaccine. Determine optimal immunogenicity of single dose in dose escalation.

In Stage 2 is to determine safety of multiple dose regimens of ShigETEC Determine number of doses for maximum immune response to Shigella and ETEC.

In both stages to determine the duration of shedding.

Stage 1 is conducted in an inpatient hospital setting at a single site through Day 6. A total of 48 subjects (2 vaccine recipients to each placebo recipient) are to be enrolled sequentially in 4 different ascending dose groups (12 subjects per group) to receive a single oral dose of the ShigETEC vaccine starting at a dose in the first group of 1 x 10^9 Colony Forming Units (CFU) of vaccine or a placebo. Each group will have baseline serum and stool samples collected at the time of admission, but in any case, before vaccination. Following 12-16 hours, they would receive oral immunization followed by evaluation of acute safety and tolerability for 6 days. Provided that no stopping rules are met through 6 days of follow-up for the entire group then the next group would be enrolled until all 4 groups were enrolled and evaluated through 6 days of assessment. Subjects in each group would be discharged to outpatient follow-up 6 days after dosing (7 days in hospital) if they were asymptomatic for shigellosis-like illness. Any subject with symptomatic illness would be treated with an appropriate course of antibiotic at the time of discharge. Daily stools will be tested for the presence of the ShigETEC vaccine until at least 2 sequential specimens are negative. If shedding persists through 14 days then the participant would be treated with antibiotics regardless of any symptomatology. All subjects would then be followed through 60 days following immunization to collect adverse events and blood samples.

Stage 2 of the study is an outpatient double-blind, placebo-controlled study. In this stage, a total of 36 subjects (2 vaccine recipients to each placebo recipient) will be enrolled in 3 different groups (12 subjects per group). The optimal dose and schedule of ShigETEC will be determined by analysis of the safety, shedding, and immunogenicity of each of the immunization schedules and interval of 3 days between doses (e.g dosing on days 1, 4, 7 and 10 for four doses.) Each group will be enrolled and followed for acute safety and tolerability from the first dose of vaccine through 6 days following the last dose of vaccine administered in their schedule and then for 60 days following the last dose of vaccine for other adverse events. Blood for serum immunogenicity studies will be obtained pre-immunization and at 6, 10, 28, and 60 days following the last immunization. Stool samples for evaluation of vaccine shedding will be collected as available (with a target of daily) through up to 14 days following the last dose of vaccine/placebo. Stool samples pre immunization and at or nearest to days 10 and 28 after the last vaccine dose for each group were evaluated for IgA titers to vaccine components. Collection of stool samples for determining vaccine shedding were terminated after two sequential negative samples after day 6 following the last dose.

ELIGIBILITY:
Inclusion Criteria:

1. Generally healthy male and non-pregnant, non-nursing female adults aged 18 to 45 years
2. Who are determined by medical history, physical examination and clinical judgment to be eligible for this study;
3. Who provide written informed consent after the nature of the study had been explained;
4. Who are available for the two to three months duration of follow-up (from enrolment to study completion);
5. Who are available to be interviewed by study staff for the 2-month post-immunization follow-up;

Exclusion Criteria:

1. Subjects who are perceived to be unavailable or difficult to contact for evaluation or study visits during the study period;
2. Who have a known or suspected disease of cancer (excluding healed skin lesions), the immune system, or those who are receiving immunosuppressive therapy, including systemic corticosteroids or cytotoxic agents;
3. Who have received any blood products, including immunoglobulin, in the period from six months prior to vaccination or are anticipated to receive such products through to the conclusion of the study;
4. Who have ever received a cholera vaccine;
5. Who are receiving antibiotics or completed antibiotic therapy in previous 7 days;
6. Who have or are participating in or have concluded participation in a clinical research study in the last 30 days or have not cleared the experimental product or the biological effects of such experimental products prior to vaccination or received a licensed vaccine in the 30 days prior to vaccination;
7. Who have a chronic non-gastrointestinal medical condition (e.g. hypertension, hyperlipidemia) that is not well controlled with medication;
8. Who have a significant history of or current diagnosis of diseases of the gastrointestinal tract (i.e. liver, gallbladder, bowel, or stomach), are on medication for such disease, or have had significant bowel surgery (with the exclusion of hernia repair or appendectomy);
9. Who have significant abnormality of blood chemistry, hematology, or screening tests (including tests for hepatitis B, HIV, HCV);
10. Who have a history of reactive arthritis following GI infection;
11. Who expect to work in the subsequent 2 weeks as a food handler or in direct patient, child day care, or elder care;
12. Who have immunocompromised household member;
13. Who have ever had a diagnosed Shigella or ETEC infection;
14. Who have developed symptoms of Shigella or ETEC infections after having travelled to Shigella or ETEC endemic areas in the past 12 months;
15. Who have any condition which in the opinion of the investigator puts the subject at risk of non-compliance with the protocol;
16. Who have known allergy to quinolone or azithromycin that will be used in the study;
17. Who are HLA-B27 positive (a possible risk factor for reactive arthritis following naturally acquired bacterial gastrointestinal infection).
18. Who are dependent of the Sponsor, of the investigational team or his/her immediate family, or are medical students at the Clinical Trial Study Site in Debrecen.
19. Who are living in community (i.e. students living in a dormitory).
20. Who are positive for CoVID19 infection by PCR testing prior to randomization.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2020-09-16 (Actual); Primary Completion 2021-06-21 (Actual); Study Completion 2021-06-21 (Actual)

PRIMARY OUTCOMES:
Number and percentage of participants with treatment related acute adverse events post vaccination | Day 1-6 following each vaccination
  Acute gastrointestinal and systemic illness symptoms following immunization(s)- treatment related Adverse events according to CTCAE v4.0 including nausea, vomiting, diarrhoea, abdominal pain, fever, joint ache, muscle/joint aches, fatigue/malaise, headache, loss of appetite.
Number and percentage of participants with any adverse event. | until 60 days after the last vaccination (max 60 days in stage 1)
  Number and percentage of participants with adverse event according to CTCAE v4.0 occuring during the entire study period
Number and percentage of participants with any adverse event. | until 60 days after the last vaccination (max 110 days in stage 2)
  Number and percentage of participants with adverse event according to CTCAE v4.0 occuring during the entire study period
Number and percentage of participants with serious adverse event. | until 60 days after the last vaccination (max 60 days in stage 1)
  Number and percentage of participants with serious adverse event occurring during the entire study period in stage 1
Number and percentage of participants with serious adverse event. | until 60 days after the last vaccination (max 110 days in stage 2)
  Number and percentage of participants with serious adverse event occurring during the entire study period in stage 2
Number and percentage of participants with Vaccine Shedding | 14 days after last immunization
  Fecal shedding of vaccine - duration of detectable presence of ShigETEC in stool by polymerase chain reaction (PCR) and/or culture.
Reactogenicity | Days 0 to 6
  Reactogenicity events accumulated through day 6 for acute safety and tolerability in acute changes in reactogenicity events at a scale (none or mild or moderate or severe) or an absolute value:
  * Temperature: degrees Celsius (°C)
  * Nausea: none/mild/moderate/severe
  * Vomiting: none/mild/moderate/severe
  * Diarrhea: none/mild/moderate/severe
  * Number of stools: discrete value
  * Abdominal pain: none/mild/moderate/severe
  * Muscle/joint aches: none/mild/moderate/severe
  * Tiredness/fatigue/malaise: none/mild/moderate/severe
  * Headache: none/mild/moderate/severe
  * Loss of appetite: none/mild/moderate/severe
  * Chills: none/mild/moderate/severe
  * Difficulty sleeping: none/mild/moderate/severe
  * Dizziness: none/mild/moderate/severe
  * Difficulty swallowing: none/mild/moderate/severe

SECONDARY OUTCOMES:
Immunogenicity assessment - serum | Day 0 and days 6, 10, 28, 60 after the last vaccination
  Serum IgA and IgG response to ShigETEC lysate, LTB and ST by ELISA
Immunogenicity assessment - ALS | Day 0 and days 6, 10 after the last vaccination
  ALS IgA response to ShigETEC lysate, LTB and ST by ELISA
Immunogenicity assessment - stool extract | Day 0 and days 10, 28 after the last vaccination
  Fecal IgA response to ShigETEC lysate, LTB and ST by ELISA; Fecal total IgA content by ELISA

CONTACTS AND LOCATIONS:
Overall Officials: Dénes Páll, MD, PhD, Principal Investigator — University of Debrecen
Locations (1):
- Debreceni Egyetem, Klinikai Központ, Belgyógyászati Klinika, Klinikai Farmakológiai Részleg, Debrecen, Hungary

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Harutyunyan S, Neuhauser I, Mayer A, Aichinger M, Szijarto V, Nagy G, Nagy E, Girardi P, Malinoski FJ, Henics T. Characterization of ShigETEC, a Novel Live Attenuated Combined Vaccine against Shigellae and ETEC. Vaccines (Basel). 2020 Nov 16;8(4):689. doi: 10.3390/vaccines8040689. PMID 33207794